CLINICAL TRIAL: NCT03118310
Title: Treatment of NAFLD With Two Different Diets
Acronym: TREND
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Hannes Hagström, Primary Investigator, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dnr 2017/258-31
Record Dates: First submitted 2017-04-06; First posted 2017-04-18 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: NAFLD
Keywords: Reduction of liver fat
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo diet
  Interventions: Behavioral: Placebo diet
- 5:2 (Experimental): 5:2 diet
  Interventions: Behavioral: 5:2 diet
- LCHF (Experimental): LCHF diet
  Interventions: Behavioral: LCHF

INTERVENTIONS:
Behavioral: 5:2 diet — Dietary intervention according to 5:2 diet during three months.
  Arms: 5:2
Behavioral: LCHF — Dietary intervention according to LCHF diet during three months.
  Arms: LCHF
Behavioral: Placebo diet — Placebo diet: normal dietary advice
  Arms: Placebo

SUMMARY:
The impact of popular diets on liver-related health is unclear. In this randomized, controlled trial, patients with NAFLD will be randomized to one of two popular diets or a placebo diet.

DETAILED DESCRIPTION:
Subjects will include patients with MRI-verified NAFLD, with no concurrent liver diseases. Randomization will be done to either a control diet, the 5:2 diet or a low-carb-high-fat diet. The subjects will follow the diet for three months, after which a new MRI is performed. Main outcomes measure is reduction in liver fat.

ELIGIBILITY:
Inclusion Criteria:

* Known NAFLD

Exclusion Criteria:

* Other forms of liver disease
* Bolus insulin treatment
* Cirrhosis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Liver fat | Three months
  MRI-measured liver fat content

CONTACTS AND LOCATIONS:
Overall Officials: Hannes Hagström, MD, PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Center for Digestive Diseases, Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holmer M, Hagstrom H, Tillander V, Alkadri M, Petersson S, Brismar TB, Stal P, Lindqvist C. One-year follow-up of short-term dietary intervention for MASLD: sustained improvements in steatosis, weight and dietary intake. Scand J Gastroenterol. 2025 Nov;60(11):1087-1095. doi: 10.1080/00365521.2025.2544305. Epub 2025 Aug 12. PMID 40797298
- [Derived] Holmer M, Lindqvist C, Petersson S, Moshtaghi-Svensson J, Tillander V, Brismar TB, Hagstrom H, Stal P. Treatment of NAFLD with intermittent calorie restriction or low-carb high-fat diet - a randomised controlled trial. JHEP Rep. 2021 Feb 17;3(3):100256. doi: 10.1016/j.jhepr.2021.100256. eCollection 2021 Jun. PMID 33898960